CLINICAL TRIAL: NCT06409039
Title: STUDIO POLE-END REAL LIFE: Carcinoma Dell'Endometrio Stadi Precoci I-II e Avanzati III e IV Valutazione di POLE Come Fattore Prognostico
Brief Title: POLE-END REAL LIFE: Endometrial Cancer Early Stages I-II and Advanced Stages III and IV Evaluation of POLE as a Prognostic Factor. Participants Are Women >= 18 Years Old, With the Pole Mutation
Acronym: POLE-END
Status: Enrolling by invitation | Type: Observational
Sponsor: Azienda Ulss 2 Marca Trevigiana (Other)
Responsible Party: Principal Investigator, Artioli Grazia, PRINCIPAL INVESTIGATOR, Azienda Ulss 2 Marca Trevigiana
Other Study IDs: GRAZIA ARTIOLI
Record Dates: First submitted 2024-04-24; First posted 2024-05-10 (Actual); Last update posted 2024-05-10 (Actual); Status verified 2024-05

CONDITIONS: Endometrial Neoplasms
MeSH Terms: conditions — Endometrial Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
POLE-END is a non-profit, observational, retrospective and prospective study which aims to analyze the clinical course of patients with POLE-mutated endometrial cancer with evaluation of Recurrence-Free Survival (RFS), defined as the interval of time between the diagnosis of POLE-mutated endometrial carcinoma and the diagnosis of disease recurrence (radiological and/or clinical and/or histological diagnosis). In particular, the investigator want to study the influence of the POLE mutation on the survival of patients and therefore on the appearance of relapses by collecting only clinical and anatomopathological-molecular data.

The study also has the secondary objective of correlating the clinical outcome with known prognostic factors and with the treatments administered.

The data will be collected on a specific Data Collection Form, made anonymous and sent to the promoting center for final analysis.

The study will be conducted according to the attached protocol, in compliance with the rules of Good Clinical Practice.

The treatment of patients will take place according to normal clinical practice and there are no additional costs borne by the Company and the Regional Health Service. Patient enrollment will take place within the centers belonging to the MITO group that have signed up.

Patients will be followed in their respective centers for the duration of their treatments and up to the fifth year after the initial diagnosis of endometrial cancer. The number of patients enrolled for this study will be approximately 80 and will have a maximum overall duration of 9 years.

As a non-profit studio, we request exemption from paying research evaluation costs.

DETAILED DESCRIPTION:
The molecular classification of endometrial carcinoma and the resulting studies have contributed to the recent ESGO/ESTRO/ESP guidelines for the management of patients diagnosed with endometrial carcinoma . To date, however, this molecular classification has mostly been performed in the context of clinical trials or in retrospective research contexts and is only now beginning to be implemented in the clinical workflow.

Endometrial carcinomas with pathogenic mutations of the POLE gene have demonstrated an excellent clinical outcome in terms of RFS and OS in the early stages of the disease (stage I and II), especially in high-grade carcinomas. Furthermore, 3-5% of endometrial carcinomas present multiple molecular alterations. In particular, the literature suggests that POLE-mutated cases that are at the same time TP53-mutated or MMR-deficient have a clinical behavior like cases with only POLE alteration. Overall, POLE-mutated tumors would therefore not require adjuvant therapy unlike carcinomas belonging to other molecular groups (TP53-mutated, MMRd and NSMP) or which are attributable to the intermediate-high risk group according to the guidelines . The PORTEC-4A study is also underway for this group.In a cohort of 23 POLE-mutated endometrial carcinomas Stasenko and colleagues documented recurrence in 17% of cases, suggesting caution in omitting adjuvant therapy. A very recent work on 310 endometrial carcinomas studied from a morpho-molecular perspective, including 15 POLE-mutated tumors, however has follow-up data that are too short to be conclusive (11.6 months on average). Advanced stage POLE-mutated carcinomas (III-IVA) are also rare and poorly described in the literature. It therefore seems appropriate to prospectively collect real-world clinical-pathological data on a large scale from patients with POLE-mutated tumors with the aim of investigating the histo-molecular characteristics of patients who undergo relapse and being able to compare them with those of non-relapsed patients. relapse. The relative rarity of POLE-mutated tumors in general and in particular of those that relapse suggests the need to involve multiple centers in order to obtain a significant number.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged > 18 years;
* Histological diagnosis of POLE-mutated endometrial carcinoma who turned to a center participating in the study starting from 01.01.2020;
* Clinical Diagnosis performed locally at each participating center including histology, immunohistochemistry and molecular evaluation;
* Signing of the informed consent to participate in the study and consent to the processing of personal data.

Exclusion Criteria:

* Patients with endometrial cancer without POLE mutation.
* Patients whose POLE status has been assessed by other methods.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Female
Study Population: Female Patients aged > 18 years with histological diagnosis of POLE-mutated endometrial carcinoma who turned to a center participating in the study starting from 01.01.2020.
  Diagnosis performed locally at each participating center including histology, immunohistochemistry and molecular evaluation.
Sampling Method: Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2023-09-04 (Actual); Primary Completion 2024-03-01 (Actual); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
POLE-END REAL LIFE STUDY: endometrial cancer early stages I-II and advanced stages III and IV evaluation of POLE as a prognostic factor | 10 years
  Recurrence-Free Survival (RFS) defined as the time interval between the diagnosis of POLE-mutated endometrial carcinoma and the diagnosis of disease recurrence (radiological and/or clinical and/or histological diagnosis),The RFS will be calculated with the Kaplan-Meier method and the 3- and 5-year values will be reported with their 95% confidence intervals, Follow-up data will be collected 3 and 5 years after diagnosis of endometrial cancer,the results will be described by means, medians, standard deviations and interquartile ranges if relating to quantitative variables and by absolute and relative frequencies for qualitative variables.

CONTACTS AND LOCATIONS:
Overall Officials: GRAZIA ARTIOLI, Principal Investigator — AULSS2 MARCA TREVIGIANA
Locations (2):
- Italy (2):
  - Aulss2 Marca Trevigiana Ospedale Ca Foncello, Treviso, TV
  - Aulss2 Marca Trevigiana Ospedale Ca Foncello, Treviso, Veneto

IPD SHARING:
Plan to Share IPD: Undecided